CLINICAL TRIAL: NCT05744180
Title: Pragmatic Analysis of the Impact and Utilization of Workflow-Integrated Artificial Intelligence for RPM Enrollment
Brief Title: A Study of Workflow-Integrated Artificial Intelligence for RPM Enrollment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tufia C. Haddad, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-008014
Record Dates: First submitted 2023-02-02; First posted 2023-02-24 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Nursing
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm Not Applicable (Other)
  Interventions: Other: Interventional

INTERVENTIONS:
Other: Interventional — The FitScore is a machine learning algorithm embedded within the electronic health record that identifies patients most likely to benefit from remote patient monitoring.
  Other Names: FitScore

SUMMARY:
The objective of this study is to evaluate effectiveness, usability and clinical utility of the remote patient monitoring (RPM) "fit" score when choosing patients to enter the RPM Program.

ELIGIBILITY:
Inclusion Criteria:

* The study participants will be nurses who are part of the RPM care team that cares for adult patients ≥18 years.
* A patient's data will be included in the analysis if the patient is ≥18 years old and receives care from a participating nurse.
* Patient data will only be collected if permitted (based on the use of the Minnesota Research Authorization Retrieval Tool).
* Patients who will be considered for this study will be assessed based on standard RPM program inclusion and exclusion criteria for the any of the chronic disease RPM programs (congestive heart failure, coronary artery disease, hypertension, type 2 diabetes, COPD, and general complex care).

Exclusion Criteria:

- < 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effectiveness, usability, and clinical utility of the RPM "fit" score as displayed in the Acute Multipatient Viewer (AMP) and underlying AI models in the real-world setting | 1 year
  FitScore effectiveness will determined by the patient care utilization outcomes of those who did or did not participate in RPM (for those enrolled with or without the FitScore). Usability and clinical utility will be self-reported by nursing staff collected through surveys or as directly observed by study staff (as to experience with or without the FitScore).

SECONDARY OUTCOMES:
Assessment of "fit" score overall effect on nursing efficiency and clinical workflows | 1 year
  Efficiency will be measured by timing studies of nurse patient screening for RPM eligibility as directly observed by study staff. The effect on clinical workflows will be self-reported by nursing staff collected through surveys (as to experience with or without the FitScore).

CONTACTS AND LOCATIONS:
Overall Officials: Tufia Haddad, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials